CLINICAL TRIAL: NCT07337252
Title: Risk Factors for the Failure of Combined Pharmacotherapy in Women With Refractory Detrusor Overactivity
Brief Title: Risk Factors for Treatment Failure in Women With Detrusor Overactivity Receiving Combined Pharmacotherapy
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Hsuan Lau, MD, Head of urogynecology, Associate Professor, Mackay Memorial Hospital
Other Study IDs: 22MMHIS039e-4
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder
Keywords: Antimuscarinic; β-agonist; Overactive Bladder; Risk factors; Treatment
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Women with urodynamic DO refractory to combined pharmacotherapy: We enrolled women with refractory detrusor overactivity, defined as ongoing symptoms after at least 1 month of treatment with either an anticholinergic or a β3-agonist. Eligible women received combined pharmacotherapy with oral solifenacin 5 mg and mirabegron 25 mg once daily for 12 weeks.
  Interventions: Drug: Combined pharmacotherapy

INTERVENTIONS:
Drug: Combined pharmacotherapy — Combined pharmacotherapy with oral solifenacin 5 mg and mirabegron 25 mg once daily.

SUMMARY:
This study evaluated the outcomes of women with detrusor overactivity treated with combined pharmacotherapy to identify risk factors for treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detrusor overactivity which defined as a urodynamic observation characterized by involuntary detrusor contractions during the filling phase. Those who were refractory to monotherapy with either anticholinergics or β3-agonist medication for at least 1 month.

Exclusion Criteria:

* Neurological conditions or spinal cord injury, which could affect urologic function
* Advanced pelvic organ prolapse (pelvic organ prolapse quantification system stage II or above)
* Active urinary tract infection
* Contraindications to taking anticholinergic and β3-agonist medications

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study focus on female overactive bladder.
Study Population: This study conducted in a tertiary referral hospital located in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Short form of Urinary Distress Inventory (UDI-6) | Assess before treatment and 12 weeks after treatment
  UDI-6 is a valid questionnaire, used particularly to investigate symptoms associated with lower urinary tract dysfunction and inquire on irritative, stress, and obstructive or discomfort complaints. UDI-6 consists of six items: frequent urination; leakage related to feeling of urgency; leakage related to activity, coughing, or sneezing; small amounts of leakage (drops); difficulty emptying the bladder; and pain or discomfort in the lower abdominal or genital area. The total score ranges from 0 to 18 , with a higher score indicating more severe of incontinence.
Short form of Incontinence Impact Questionnaire (IIQ-7) | Assess before treatment and 12 weeks after treatment
  The IIQ-7 assess the impact of urinary incontinence on QoL. 7 items assess influence of urinary incontinence on physical activity, travel, social/relationships & emotional health. Each item is scored between 0 (activities not affected at all) to 3 (activities greatly affected). The total score ranges from 0 to 21, with a higher score indicating more severe of incontinence.
Overactive Bladder Symptom Score (OABSS) | Assess before treatment and 12 weeks after treatment
  The total OABSS is the sum of four symptom scores: daytime frequency (score 0-2), nighttime frequency (score 0-3), urgency (score 0-5), and urgency incontinence (score 0-5). The total score ranges from 0 to 15, with a higher score indicating more severe of OAB symptoms.

SECONDARY OUTCOMES:
Episodes of daily micturition | Assess before treatment and 12 weeks after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily urgency | Assess before treatment and 12 weeks after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily incontinence | Assess before treatment and 12 weeks after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily nocturia | Assess before treatment and 12 weeks after treatment
  Patients report daily lower urinary tract symptoms episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No